CLINICAL TRIAL: NCT07101874
Title: A Retrospective Study of Biliary Complications and Treatment Duration in Patients With Biliary Tract Cancer Receiving Systemic Therapy in Japan
Brief Title: A Study to Evaluate the Association of Biliary Complications and Treatment Duration in Unresectable BTC Patients
Acronym: ARCBile
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Japan Oncology Network in Hepatobiliary and Pancreas (JON-HBP) (Unknown)
Responsible Party: Sponsor
Other Study IDs: D4191R00099
Record Dates: First submitted 2025-06-10; First posted 2025-08-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This is a multi-center, retrospective, observational study of patients receiving first-line systemic therapy as routine clinical care for unresectable BTC in Japan. This study attempts to test the hypothesis that the occurrence of biliary complications requiring hospitalization during first-line systemic therapy for unresectable BTC, which is as a time-dependent covariate, affects time to treatment failure (TTF) .

DETAILED DESCRIPTION:
The real-world evidence on cancer-related biliary complications during systemic therapy in patients with advanced biliary tract cancers (BTC) in a large population is lacking. The results from this study may reveal the association of biliary complications with treatment duration, provide an overview of the current status of managing them, and clarify the issues to be addressed as a priority in future studies.

This is a multi-center, retrospective, observational study of patients receiving first-line systemic therapy as routine clinical care for unresectable BTC in Japan.

The primary objective of this study is to evaluate the association of the occurrence of biliary complication during first-line systemic therapy with time to treatment failure (TTF) in unresectable BTC patients, to test the hypothesis that the occurrence of biliary complications requiring hospitalization during first-line systemic therapy for unresectable BTC as a time-dependent covariate is significantly associated with TTF .

This study is conducted in collaboration with Japan Oncology Network in Hepatobiliary and Pancreas (JON-HBP, https://jon-hbp.org/en/). Approximately 1,000 patients who start the first dose of first-line systemic therapy for unresectable BTC between May 1, 2022, and December 31, 2023, will be enrolled and these patients' data until July 31, 2025 in medical charts will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with "unresectable BTC" who meet any of the following:

1. Patients who were deemed unamenable to curative resection at the initial diagnosis.
2. Patients who relapsed after curative resection of BTC more than 6 months after the end of adjuvant therapy or after the date of surgery for patients who did not receive adjuvant therapy.

2. Patients who received first-line systemic therapy for unresectable BTC with the date of the first dose between May 1, 2022, and December 31, 2023. However, patients who received postoperative adjuvant therapy for BTC with R2 resection is not included.

3. Patients with ECOG performance status 0 or 1 on the most recent assessment date prior to first dose of first-line systemic therapy for unresectable BTC 4. Patients who provided written informed consent form (ICF), in cases where obtaining informed consent is not difficult, or for whom an appropriate opt-out approach was taken at the study site if obtaining informed consent is difficult.

5. Patients aged 18 years or older at the date of first dose of first-line systemic therapy for unresectable BTC.

6. Patients who started first-line systemic therapy with physician's expectation of 3 months or longer prognosis at the time of starting systemic therapy.

Exclusion Criteria:

1. Maintenance dialysis at the date of the first dose of first-line systemic therapy for unresectable BTC.
2. Combined any locoregional therapy with first-line systemic therapy for unresectable BTC (e.g., radiation therapy, radiofrequency ablation, arterial injection chemotherapy)
3. Patient who participated in clinical trials (interventional studies) of first-line systemic therapy for BTC
4. Active cancers other than unresectable BTC within the past 2 years from the date of the first dose of first-line systemic therapy. The following are exceptions to this criterion:

   * Carcinoma in situ or lesions equivalent to carcinoma in situ.
   * Intramucosal cancers that are deemed cured by local treatment.
5. Patients who were followed up for less than 3 months after starting first-line systemic therapy for reasons other than TTF events (disease progression, death, or treatment discontinuation).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of approximately 1,000 patients who received first-line systemic therapy for unresectable BTC including intrahepatic/perihilar/distal cholangiocarcinoma, GBC, or cancer of the AoV will be the study population. And in this study, the patients with unresectable BTC were defined as follows:
  1. Patients who were deemed unamenable to curative resection at the initial diagnosis.
  2. Patients who relapsed after curative resection of BTC more than 6 months after the end of adjuvant therapy or after the date of surgery for patients who did not receive adjuvant therapy.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure (TTF) | From 1st dose of first-line systemic therapy until disease progression or death by any cause or discontinuation of first-line systemic therapy for unresectable BTC by physician's decision, whichever came first, assessed up to 2 years.
  TTF is defined as the time from the first dose date of first-line systemic therapy to the earliest date of any following events;
  1. Disease progression determined by physicians.
  2. Death by any cause.
  3. Discontinuation of first-line systemic therapy for unresectable BTC by physician's decision.
  The impact of biliary complications on first-line systemic therapy will be evaluated by HR with 95% confidence interval (CI) which is estimated with TTF and incidence rate of event in the patient group who developed biliary complication before a certain time t and patient group who did not develop biliary complication before time t.

SECONDARY OUTCOMES:
The number and proportion of patients with each reason for discontinuation (including disease progression and cause of death) of first-line systemic therapy. | From 1st dose of first-line systemic therapy until disease progression or death by any cause or discontinuation of first-line systemic therapy for unresectable BTC by physician's decision, whichever came first, assessed up to 2 years.
  Patient group:
  1. Overall study population.
  2. Patient group with/without pre-treatment biliary drainage before starting first-line systemic therapy within overall study population.
The number and proportion of patients per the number (including zero) of occurrence of biliary complications during first-line systemic therapy. | From 1st dose of first-line systemic therapy until disease progression or death by any cause or discontinuation of first-line systemic therapy for unresectable BTC by physician's decision, whichever came first, assessed up to 2 years.
  Patient group:
  1. Overall study population.
  2. Patient group with/without pre-treatment biliary drainage before starting first-line systemic therapy within overall study population.
The detail following information of the first biliary complication during first-line systemic therapy, e.g., Disease classification, Bacteremia, Main site of obstruction or stenosis. | The duration of hospitalization due to the first biliary complication requiring admission up to July 31, 2025.
  All information related the first biliary complication.

CONTACTS AND LOCATIONS:
Locations (22):
- Japan (22):
  - Research Site, Aichi
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kyoto
  - Research Site, Miyagi
  - Research Site, Nara
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saitama
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokyo
  - Research Site, Wakayama

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to de-identified individual patient-level data from AstraZeneca group of companies sponsored clinical trials/studies via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://vivli.org/